CLINICAL TRIAL: NCT06796283
Title: Research on AIS Recurrence Risk Prediction Model Using XGBoost Combined With Convolutional Neural Network Algorithm
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021efyB03
Record Dates: First submitted 2025-01-13; First posted 2025-01-28 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this observational study is to construct a recurrence risk prediction model for ischemic stroke within 1, 3, 6, and 12 months using XGBoost combined with Convolutional Neural Network (CNN) algorithm.

Method: Follow up was conducted on the study subjects at 1, 3, 6, and 12 months after discharge.

Follow up primary outcome: Whether the study subjects experienced recurrent stroke events.

Secondary outcome: Improved Rinkin score.

Collect information on research subjects:

It includes demographic data, physical examination, medical history, imaging images, medication use, scale scores, CYP2C19 genotype test results, laboratory tests, and other complex multidimensional data.

DETAILED DESCRIPTION:
This project conducts a one-year follow-up on the enrolled subjects (patients with ischemic stroke) to observe the recurrence and modified Rankin scores after discharge. Combining complex multidimensional data such as demographic information, physical examination, medical history, imaging images, medication status, NIHSS scale scores, Glasgow Coma Scale scores, CYP2C19 genotype test results, and laboratory examinations of the subjects; Convolutional Neural Networks (CNNs) are used to segment lesions and extract features from the subjects' imaging images; Cox regression models are employed to obtain factors influencing recurrence; a prediction model for the risk of recurrence within 1, 3, 6, and 12 months for ischemic stroke is constructed using the XGBoost algorithm combined with Convolutional Neural Networks. The exploration aims to provide new insights and methods for the prevention and control of major chronic diseases by evaluating the effectiveness of XGBoost in predicting the risk of ischemic stroke recurrence at different times.

1. Inclusion Criteria：

   * 18-85 years old;
   * Diagnosed with ischemic stroke or transient ischemic attack (diagnosis meets the criteria established by the Cerebrovascular Disease Group of the Neurology Branch of the Chinese Medical Association in 2014);
   * During the acute phase of onset (2 weeks);
   * Voluntarily participate and sign an informed consent form.
2. Exclusion criteria：

   * Cancer patients;
   * Cardiogenic infarction, cerebral infarction of other causes, and cerebral infarction of unknown causes;
   * Patients with hemorrhagic stroke, mixed stroke, and tumor stroke;
   * Merge with severe heart, lung, and liver system diseases;
   * Researchers identify patients with poor compliance and inability to complete long-term follow-up;
   * Patients currently participating in any clinical trials related to investigational drugs or medical devices.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-85 years
* Diagnosed with ischemic stroke or transient ischemic attack (diagnosis in accordance with the standards set by the Cerebrovascular Disease Group of the Neurology Branch of the Chinese Medical Association in 2014)
* Within the acute phase of the illness (within 2 weeks)
* Voluntarily participates and signs an informed consent form

Exclusion Criteria:

* Patients with cancer
* Patients with cardiogenic infarction, other causes of cerebral infarction, or cryptogenic cerebral infarction
* Patients with hemorrhagic stroke, mixed stroke, and tumor stroke
* Patients with severe heart, lung, or liver system diseases
* Patients judged by the researcher to have poor compliance and unable to complete long-term follow-up
* Patients currently participating in any clinical trials related to investigational drugs or medical devices

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke patients treated in hospitals who meet the inclusion and exclusion criteria for the project
Sampling Method: Non-Probability Sample
Enrollment: 2628 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrent ischemic stroke, | April 6th, 2021- March 12th, 2024
  Follow up was conducted on the study subjects at 1, 3, 6, and 12 months after discharge, with the main outcome being whether the study subjects experienced stroke recurrence events

SECONDARY OUTCOMES:
modified Rankin score | April 6th, 2021- March 12th, 2024
  Follow up was conducted on the study subjects at 1, 3, 6, and 12 months after discharge, with the secondary outcome being the modified Rinkin score.Improved Rinkin Scale:
  Completely asymptomatic (0 points). Despite symptoms, there is no obvious functional impairment and the ability to complete all daily work and life tasks (1 point).
  Mild disability, unable to complete all pre illness activities, but able to take care of daily affairs without assistance (2 points).
  Moderate disability, requiring partial assistance, but able to walk independently (3 points).
  Moderate to severe disability, unable to walk independently, requiring assistance from others in daily life (4 points).
  Severe disability, bedridden, urinary incontinence, and complete dependence on others in daily life (5 points).
  The higher the score, the worse the participant's neurological function recovery.

CONTACTS AND LOCATIONS:
Overall Officials: yingping Y Yi, Principal Investigator — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu J, Li J, Wu Y, Luo H, Yu P, Cheng R, Wang X, Xian H, Wu B, Chen Y, Ke J, Yi Y. Deep learning-based segmentation of acute ischemic stroke MRI lesions and recurrence prediction within 1 year after discharge: A multicenter study. Neuroscience. 2025 Jan 26;565:222-231. doi: 10.1016/j.neuroscience.2024.12.002. Epub 2024 Dec 2. PMID 39631660
- See also: Explore deep - learning - based infarct lesion segmentation in AIS patients' brain MRI, radiomics - based 1 - year recurrence prediction, and develop a combined model for accurate AIS recurrence prediction — https://pubmed.ncbi.nlm.nih.gov/39631660/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT06796283/Prot_SAP_ICF_000.pdf